CLINICAL TRIAL: NCT04253743
Title: Evaluation of Demonstrations to End Childhood Hunger - Nevada
Brief Title: Evaluation of Demonstrations to End Childhood Hunger - NV
Acronym: EDECHNV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA Food and Nutrition Service (U.S. Federal Agency)
Collaborators: Mathematica Policy Research, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AG-3198-C-14-0019 (Nevada)
Record Dates: First submitted 2019-12-12; First posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Food Insecurity Among Children
Keywords: Food security; Hunger; Young children; Supplemental Nutrition Assistance Program (SNAP); Food expenditures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nevada Healthy, Hunger-Free Kids Demonstration Benefits (Experimental): SNAP households were randomly assigned to receive either: (1) $40 extra in SNAP benefits per eligible child (<5 years) per month (n=1,919); (2) $40 extra in SNAP benefits per eligible child per month plus case management and nutrition education (n=1,919); or (3) only regular monthly SNAP benefit (n=7,467). The first two groups were the treatment arms and the third was the control group.
  Interventions: Other: Nevada Healthy, Hunger-Free Kids Demonstration Benefits
- Control Group (No Intervention): The control group received regularly allotted SNAP benefits.

INTERVENTIONS:
Other: Nevada Healthy, Hunger-Free Kids Demonstration Benefits — SNAP households with children under age 5 incomes below 75% of the federal poverty level living in Clark County, Nevada received $40 in extra SNAP benefits per eligible child, and access to case management and nutrition education.
  Arms: Nevada Healthy, Hunger-Free Kids Demonstration Benefits

SUMMARY:
The 2010 Child Nutrition Reauthorization provided funding to test innovative strategies to end childhood hunger and food insecurity. Demonstration projects were funded in Chickasaw Nation, Kentucky, Navajo Nation, Nevada, and Virginia. This study focuses on Nevada.

SNAP households were randomly assigned to receive either: (1) $40 extra in SNAP benefits per eligible child (<5 years) per month; (2) $40 extra in SNAP benefits per eligible child per month plus case management and nutrition education; or (3) only regular monthly SNAP benefit. The first two groups were the treatment arms and the third was the control group.

DETAILED DESCRIPTION:
Objectives: To (1) reduce food insecurity among children; (2) increase enrollment in the Special Supplemental Nutrition Program for Women, Infants, and Children (WIC) and other nutrition assistance programs; and (3) improve nutrition and healthy shopping habits through nutrition education.

Target Population: Supplemental Nutrition Assistance Program (SNAP) households with children under age 5 and incomes below 75 percent of the Federal Poverty Level living in Clark County, Las Vegas, Nevada.

Intervention: SNAP households were randomly assigned to receive either: (1) $40 extra in SNAP benefits per eligible child (<5 years) per month; (2) $40 extra in SNAP benefits per eligible child per month plus case management and nutrition education; or (3) only regular monthly SNAP benefit. The first two groups were the treatment arms and the third was the control group.

The two treatment groups were ultimately combined because of the low uptake of case management and nutrition education.

ELIGIBILITY:
Inclusion Criteria:

* Supplemental Nutrition Assistance Program (SNAP) households with children under age 5 and incomes below 75 percent of the Federal Poverty Level living in Clark County, Las Vegas, Nevada.

Max Age: 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 7246 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Food Insecurity among Children | 30 days
  Measured by the United States Department of Agriculture's Household Food Security Survey Module (HFSSM).
  Affirming 2 or more out of the 8 child-level items in the HFSSM. Higher scores generally indicates worsening food insecurity.

SECONDARY OUTCOMES:
Very Low Food Insecurity among Children | 30 days
  Measured by the United States Department of Agriculture's Household Food Security Survey Module (HFSSM).
  Affirming 5 or more out of the 8 child-level items in the HFSSM. Higher scores generally indicates worsening food insecurity.
Food Insecurity among Adults | 30 days
  Measured by the United States Department of Agriculture's Household Food Security Survey Module (HFSSM).
  Affirming 3 or more out of the 10 adult-level items in the HFSSM. Higher scores generally indicates worsening food insecurity.
Household Food Insecurity | 30 days
  Measured by the United States Department of Agriculture's Household Food Security Survey Module (HFSSM).
  Affirming 3 or more out of the 18 items in the HFSSM. Higher scores generally indicates worsening food insecurity.
Food Expenditures | 30 days
  Total amount of Supplemental Nutrition Assistance Program (SNAP) and out-of-pocket food purchases in dollars

CONTACTS AND LOCATIONS:
Overall Officials: Michael P Burke, PhD, Study Director — USDA Food and Nutrition Service

IPD SHARING:
Plan to Share IPD: Yes
Public-use data files are available by request by contacting Michael Burke (michael.burke@usda.gov) or the Office of Policy Support within the USDA Food and Nutrition Service.
Time Frame: April 2019

REFERENCES:
- [Derived] Gleason PM, Kleinman R, Chojnacki GJ, Briefel RR, Forrestal SG. Measuring the Effects of a Demonstration to Reduce Childhood Food Insecurity: A Randomized Controlled Trial of the Nevada Healthy, Hunger Free Kids Project. J Acad Nutr Diet. 2021 Jan;121(1S):S22-S33. doi: 10.1016/j.jand.2020.03.002. PMID 33342522
- See also: Final Report — https://www.fns.usda.gov/ops/evaluation-demonstration-projects-ech